CLINICAL TRIAL: NCT02410044
Title: Open-labeled, Multicenter, Non-interventional Prospective PRO/QoL Registry for Patients With Osteoprotective Treatment for Bone Metastases of Breast or Prostate Cancer
Brief Title: Prospective PRO/QoL Registry for Patients With Bone Metastases of Breast or Prostate Cancer
Acronym: PROBone
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM - 11279
Record Dates: First submitted 2014-12-23; First posted 2015-04-07 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Prostate Cancer; Bone Metastases
Keywords: Patient Reported Outcomes
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of patient reported outcomes (PRO) / QoL regarding typical ailments in real-life patients with bone metastases treated with osteoprotective agents.

DETAILED DESCRIPTION:
The PRO Bone project will recruit a representative cohort of patients with breast or prostate cancer suffering from bone metastases. The aim of this study is to collect data on Patient Reported Outcomes (PRO)/Quality of Life regarding bone pain and the impact of bone pain on quality of life and daily activities. PROs are assessed by a questionnaire consisting of a visual analog scale for bone pain, two questions regarding bone pain management, the bone pain module of FACT questionnaire (FACT-BP) and four questions addressing the impact of treatment on daily life (overall, social life, ability to work and ability to perform routine tasks)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast or prostate cancer
* Start of first systemic osteoprotective treatment
* Ability to read and understand German
* Written informed consent

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastasized breast or prostate cancer at the start of first systemic osteoprotective treatment for bone metastases
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-12-23 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2020-08-16 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes (PRO) regarding bone pain and the impact of bone pain on quality of life and daily activities in patients with bone metastases treated with osteoprotective agents. | 12 months

SECONDARY OUTCOMES:
Patient Reported Outcomes regarding the impact of treatment on daily life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark-Oliver Zahn, MD, Study Chair — medical practise for oncology
Locations (1):
- Multiple sites all over Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No